CLINICAL TRIAL: NCT04616066
Title: Effect of Date Fruit Phytoestrogen on the Glycemic Control of Patients With Type 2 Diabetes: A Randomized Clinical Trial.
Brief Title: Date Fruit Effects in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons in Ireland - Medical University of Bahrain (Other)
Collaborators: King Hamad University Hospital, Bahrain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 89 / 25-Oct-2020
Record Dates: First submitted 2020-10-25; First posted 2020-11-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Type2 Diabetes
Keywords: Type2 diabetes; Dates; Phytoestrogen
MeSH Terms: interventions — Chronology as Topic

STUDY DESIGN:
Intervention Model Description: This is a parallel, prospective, interventional and randomized trial involving 80 patients with type 2 diabetes. They will be randomised to either 60g of dates or 60g of raisins (amount split and given as a mid-morning and mid-afternoon snack) for 3 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dates Arm (Experimental): Consumption of Khalas dates (3 dates =30g undried dates) twice daily (phytoestrogen content 329ug/100g)
  Interventions: Other: Dates
- Raisins Arm (Experimental): Consumption of Raisins (30g twice daily, phytoestrogen content of 9.6ug/100g)
  Interventions: Other: Raisins

INTERVENTIONS:
Other: Dates — The effect of date phytoestrogens on HbA1C and fasting blood glucose in patients with type 2 diabetes
  Arms: Dates Arm
Other: Raisins — The effect of raisins phytoestrogens on HbA1C and fasting blood glucose in patients with type 2 diabetes
  Arms: Raisins Arm

SUMMARY:
Dried dates (Phoenix dactylifera) have the second highest phytoestrogen content of any fruit, only secondary to dried apricots with 329ug of phytoestrogens per 100g. The date palm is one of oldest planted trees on the earth at around 2,000 years old. Dates are nutritionally rich and a good source of fiber and carbohydrates and their potential medicinal and nutritional effects have been suggested in a number of studies. Date sugars have also been shown to be phenol rich, potent antioxidant, and strong inhibitor of α -glycosidase that may also have benefit in diabetes. In addition, dates are rich in micronutrients that may also have benefit for diabetes and insulin resistance . Dates have a glycemic index of 50 and studies have shown that the consumption of differing varieties of dates do not significantly affect the acute glycemia in patients with type 2 diabetes.

The objective of this study is to investigate the effect of date phytoestrogens on HbA1C and fasting blood glucose in patients with type 2 diabetes in comparison to the same glycemic load of raisins that have low phytoestrogen content.

DETAILED DESCRIPTION:
Production and consumption of soy foods within Western countries have increased dramatically in the last decade with the postulated health benefits including improvement in bone health, relief of menopausal symptoms and reduced risk of certain types of cancers due to the soy phytoestrogens. In addition, habitual intake of soy phytoestrogens has also been associated with a reduced risk of type 2 diabetes mellitus (T2DM) and cardiovascular disease (CVD), which is of particular relevance given the increasing global prevalence of diabetes. This is a particular problem here in the Middle East and North Africa (MENA) region, where diabetes is considered as a serious and increasing health problem. According to the International Diabetes Federation the prevalence of diabetes in the MENA region is over 23.3%; however worldwide there is an epidemic increase in type 2 diabetes with the WHO report that approximately 415 million people have diabetes worldwide, and that by 2030, diabetes will be the 7th leading cause of death.

Dried dates (Phoenix dactylifera) have the second highest phytoestrogen content of any fruit, only secondary to dried apricots with 329ug of phytoestrogens per 100g. The date palm is one of oldest planted trees on the earth at around 2,000 years old. Dates are nutritionally rich and a good source of fiber and carbohydrates and their potential medicinal and nutritional effects have been suggested in a number of studies. Date sugars have also been shown to be phenol rich, potent antioxidant, and strong inhibitor of α -glycosidase that may also have benefit in diabetes. In addition, dates are rich in micronutrients that may also have benefit for diabetes and insulin resistance. Dates have a glycemic index of 50 and studies have shown that the consumption of differing varieties of dates do not significantly affect the acute glycemia in patients with type 2 diabetes.

There has not been a medium term study of the effect of date fruit in diabetes; therefore, this study will determine if the consumption Khalas dates (3 dates =30g undried dates) twice daily (phytoestrogen content 329ug/100g), in accord with that advised in the Holy Qur'an, will improve the glycemic control in men with type 2 diabetes, in comparison with the equivalent glycemic load of raisins (30g twice daily, phytoestrogen content of 9.6ug/100g). Each intervention will be taken as a snack mid-morning and mid-afternoon.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of type 2 diabetes will be based on the WHO guidelines. An HbA1C of 6.5% or greater, or 2 fasting plasma glucose readings of >7.0mmoll-1 or 2 random plasma glucose readings >11mmoll-1 in the absence of symptoms or concurrent illness or medication which might lead to hyperglycaemia (e.g. thiazide diuretics). Or one reading meets the diagnostic level with the presence of symptoms of polyuria, polydipsia, nocturia, fatigue or blurring of vision. The final diagnostic method of diagnosis type 2 diabetes is a positive oral glucose tolerance test (OGTT) using a 75g glucose load. If doubt exists on the diagnosis of diabetes an OGTT will be performed.
* Patients will be on stable medication for their diabetes, hypertension, lipids and gout (if appropriate) for 3 months prior to entry into the study.
* HbA1c 7.5 - 10%
* Patients between the ages of 45-75 years at the start of the study.
* Capable to give informed consent and complete the study.

Exclusion Criteria:

* Patients with concurrent illness or any medication in the last 3 months.
* Patients who are taking hormone replacement therapy.
* Patients who are currently or have taken antibiotics in the last 3 months.
* Currently enrolled in other clinical trials.
* Hba1c at recruiting stage of more than 10%.
* Patients with a BMI less than 20 and more than 40.
* Patients with known food allergies.
* Patients on insulin.
* Patients who are eating dates or raisins should be washed out for 4 weeks.
* Pregnant or nursing, or plans to become pregnant in the next 3 months, or not using adequate contraceptive measures.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
The effect of phytoestrogens on HbA1C and fasting blood glucose in patients with type 2 diabetes | 90 days
  Measuring the levels of phytoestrogen and evaluate if it has reduced the average blood sugar levels over a period of 3 months.

SECONDARY OUTCOMES:
Determine whether date phytoestrogens affect cardiovascular risk | 90 days
  Determine whether the level of phytoestrogens has lowered risks of cardiovascular disease by measuring the fasting lipids, C reactive protein and blood pressure.
Determine whether date phytoestrogens affect insulin resistance | 90 days
  Homeostatic model assessment (HOMA) is a method for assessing β-cell function and insulin resistance (IR) from basal (fasting) glucose and insulin or C-peptide concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Naji Alamuddin, Dr., Principal Investigator — Royal College of Surgeons in Ireland - Bahrain
Locations (1):
- Royal College of Surgeons in Ireland - Bahrain, Manama, Bahrain

IPD SHARING:
Plan to Share IPD: Yes
Monitoring, audits, and REC review will be permitted and provide direct access to source data and documents. The Lead PI and the researchers assigned by him will have access to the stored data/specimens. Only the Lead PI and the researchers assigned working on this study will be eligible to obtain the data/specimens from the participants during data collection.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Dr Naji will act as the data custodian and is responsible for the storage, handling and quality of the study data.
  Data will be collected in the case report form to allow for cross referencing to check validity.
  Study documents (paper and electronic) will be retained in a secure (kept locked when not in use) location during and after the trial has finished. All essential documents including source documents will be retained for a period of 3 years after study completion (last patient, last study point). A label stating the date after which the documents can be destroyed will be placed on the inside front cover of the case notes of trial participants.
Access Criteria: Study documents (paper and electronic) will be retained in a secure (kept locked when not in use) location during and after the trial has finished.

REFERENCES:
- [Background] Xiao CW. Health effects of soy protein and isoflavones in humans. J Nutr. 2008 Jun;138(6):1244S-9S. doi: 10.1093/jn/138.6.1244S. PMID 18492864
- [Background] Jayagopal V, Albertazzi P, Kilpatrick ES, Howarth EM, Jennings PE, Hepburn DA, Atkin SL. Beneficial effects of soy phytoestrogen intake in postmenopausal women with type 2 diabetes. Diabetes Care. 2002 Oct;25(10):1709-14. doi: 10.2337/diacare.25.10.1709. PMID 12351466
- [Background] Xu SZ, Zeng B, Daskoulidou N, Chen GL, Atkin SL, Lukhele B. Activation of TRPC cationic channels by mercurial compounds confers the cytotoxicity of mercury exposure. Toxicol Sci. 2012 Jan;125(1):56-68. doi: 10.1093/toxsci/kfr268. Epub 2011 Oct 9. PMID 21984481
- [Background] Thompson LU, Boucher BA, Liu Z, Cotterchio M, Kreiger N. Phytoestrogen content of foods consumed in Canada, including isoflavones, lignans, and coumestan. Nutr Cancer. 2006;54(2):184-201. doi: 10.1207/s15327914nc5402_5. PMID 16898863
- [Background] Vayalil PK. Date fruits (Phoenix dactylifera Linn): an emerging medicinal food. Crit Rev Food Sci Nutr. 2012;52(3):249-71. doi: 10.1080/10408398.2010.499824. PMID 22214443
- [Background] Hamad I, AbdElgawad H, Al Jaouni S, Zinta G, Asard H, Hassan S, Hegab M, Hagagy N, Selim S. Metabolic Analysis of Various Date Palm Fruit (Phoenix dactylifera L.) Cultivars from Saudi Arabia to Assess Their Nutritional Quality. Molecules. 2015 Jul 27;20(8):13620-41. doi: 10.3390/molecules200813620. PMID 26225946
- [Background] Alkaabi JM, Al-Dabbagh B, Ahmad S, Saadi HF, Gariballa S, Ghazali MA. Glycemic indices of five varieties of dates in healthy and diabetic subjects. Nutr J. 2011 May 28;10:59. doi: 10.1186/1475-2891-10-59. PMID 21619670
- [Background] Alkaabi J, Al-Dabbagh B, Saadi H, Gariballa S, Yasin J. Effect of traditional Arabic coffee consumption on the glycemic index of Khalas dates tested in healthy and diabetic subjects. Asia Pac J Clin Nutr. 2013;22(4):565-73. doi: 10.6133/apjcn.2013.22.4.09. PMID 24231017
- [Background] Miller CJ, Dunn EV, Hashim IB. The glycaemic index of dates and date/yoghurt mixed meals. Are dates 'the candy that grows on trees'? Eur J Clin Nutr. 2003 Mar;57(3):427-30. doi: 10.1038/sj.ejcn.1601565. PMID 12627179
- [Background] Senn SJ. Covariate imbalance and random allocation in clinical trials. Stat Med. 1989 Apr;8(4):467-75. doi: 10.1002/sim.4780080410. PMID 2727470
- [Background] Senn S. Testing for baseline balance in clinical trials. Stat Med. 1994 Sep 15;13(17):1715-26. doi: 10.1002/sim.4780131703. PMID 7997705
- [Background] Knol MJ, Groenwold RH, Grobbee DE. P-values in baseline tables of randomised controlled trials are inappropriate but still common in high impact journals. Eur J Prev Cardiol. 2012 Apr;19(2):231-2. doi: 10.1177/1741826711421688. No abstract available. PMID 22512015